CLINICAL TRIAL: NCT01062048
Title: Re-examination Study for General Drug Use to Assess the Safety and Efficacy Profile of Januvia in Usual Practice
Brief Title: Januvia Re-examination Study (MK-0431-181)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0431-181; 2010_003 (Other: Merck Registration Number)
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Sulfonylurea Compounds; Insulin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Participants administered Januvia up to 100 mg once daily as monotherapy or combination therapy with a sulfonylurea or with insulin during the re-examination period (up to 6 years)
  Interventions: Drug: Sitagliptin; Drug: Sulfonylurea; Biological: Insulin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin phosphate monohydrate 25 mg, 50 mg, or 100 mg tablet administered in general use according to the local label
  Other Names: Januvia
Drug: Sulfonylurea — Sulfonylurea administered in general use according to the local label
Biological: Insulin — Insulin administered in general use according to the local label

SUMMARY:
The objectives of this survey are: 1) To examine the safety/efficacy profile of Januvia in Korean participants, and 2) To identify factors that might have an influence on the safety and efficacy profile of Januvia in Korean participants.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Treated With Januvia within local label for the first time

Exclusion Criteria:

* Contraindication to Januvia according to the local label
* Treated with Januvia before contract and out of enrollment period

Inclusion criteria for long-term surveillance

* Treated with Januvia for more than or equal to 24 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean participants with Type 2 Diabetes Mellitus being treated with Januvia
Sampling Method: Probability Sample
Enrollment: 3483 (Actual)
Dates: Start 2008-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with any adverse experience | up to 14 days following cessation of treatment
Mean change in Hemoglobin A1c (HbA1c) | 12 weeks ± 2 weeks and 24 weeks ± 2 weeks after first treatment
Mean change in fasting plasma glucose (FPG) | 12 weeks ± 2 weeks and 24 weeks ± 2 weeks after first treatment
Mean change in 2hr-postprandial glucose (PPG) | 12 weeks ± 2 weeks and 24 weeks ± 2 weeks after first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC